CLINICAL TRIAL: NCT02333266
Title: Bio-assay Development and Implementation for Fungal Infection Detection
Status: Withdrawn | Type: Observational
Why Stopped: The bioassay development is too difficult.
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Sponsor
Other Study IDs: S57146
Record Dates: First submitted 2014-12-17; First posted 2015-01-07 (Estimated); Last update posted 2016-05-12 (Estimated); Status verified 2015-12

CONDITIONS: Candidemia
Keywords: Candida bloodstream infection; Detection fungal cells; Fiber-Optic Surface Plasmon Resonance (FO-SPR)
MeSH Terms: conditions — Candidemia

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Whole blood samples
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Candidemia: 0
  Interventions: Other: Candidemia

INTERVENTIONS:
Other: Candidemia

SUMMARY:
The purpose of this study is to determine whether the newly developed biosensor can be used to detect and quantify fungal cells in human blood samples.

DETAILED DESCRIPTION:
The study discussed here is part of a broader research project (IOF project) that is aimed at the development and implementation of a point-of-care devices, in which Fiber-Optic Surface Plasmon Resonance (FO-SPR) is used as a detection system. This project includes the development and implementation of the (FUNGDETECT) sensor for fast and accurate detection of fungal pathogens in human blood samples. In first instance, the sensor will be tested in buffer solutions spiked with a known amount of Candida albicans cells. Further validation of the prototype includes detection of these cells in human blood samples. In a first experiment, detection of yeast cells will be performed in blood samples from 5 healthy volunteers each spiked with yeast cells from different Candida spp.. A second experiment includes the detection in blood samples from 15 patients who suffer from a candidemia. The blood samples will be collected from patients of University Hospitals (UZ) Leuven.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers for validation of the (FUNGDETECT) sensor (Spiked blood samples)
* Candidemia

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients laying in the hospital that suffer from a candidemia.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2016-06; Primary Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Detection of Candida albicans with the newly developed FUNGDETECT sensor in blood samples from patients with candidemia due to Candida albicans | Blood samples will be collected at baseline from patients directly after informed consent is given
  Patients in the hospital and suspected to have a Candida infection will be tested for Candida infections via blood cultures. Blood samples for patients with a positive test will be taken immediately after the positive result and used to validate the FUNGDETECT sensor.

CONTACTS AND LOCATIONS:
Overall Officials: Jeroen Lammertyn, Prof., Study Director — KU Leuven; Katrien Lagrou, Prof., Principal Investigator — Universitaire Ziekenhuizen KU Leuven